CLINICAL TRIAL: NCT06559774
Title: The Hastiin Bidziil (Strong Man) Intervention: A Study to Measure the Effectiveness of a Secondary Prevention Program Aimed at Reducing Substance Use Among Native Men Ages 18-30
Brief Title: The Hastiin Bidziil (Strong Man) Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00027710
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Substance Use
Keywords: Young Men; Common Elements Treatment Approach (CETA)
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The co-Leads (project Investigators) are blinded to randomization status of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hastiin Bidziil (Strong Man) intervention (Experimental): CETA intervention adapted for AI men ages 18-26. Adaptation will take place leading up to implementation of the randomized controlled trial
  Interventions: Behavioral: Hastiin Bidziil
- Active Control Group - Vehicle Maintenance (Placebo Comparator): Control condition was selected by the Community Research Council and includes five sessions on basic vehicle maintenance.
  Interventions: Other: Control condition - vehicle maintenance

INTERVENTIONS:
Behavioral: Hastiin Bidziil — Common Elements Treatment Approach (CETA) modified for cultural and gendered specific delivery for maximum community impact
  Arms: Hastiin Bidziil (Strong Man) intervention
Other: Control condition - vehicle maintenance — Control condition was selected by the Community Research Council and includes five sessions on basic vehicle maintenance such as changing tire, checking fluid levels, and winterizing vehicles.
  Arms: Active Control Group - Vehicle Maintenance

SUMMARY:
The Hastiin Bidziil (Strong man) Intervention study is part of a larger project called, Community-Driven Indigenous Research, Cultural Strengths & Leadership to Advance Equity in Substance Use Outcomes (CIRCLE) Center of Excellence. CIRCLE aims to address drug use related health problems in collaboration with diverse Indigenous communities. This study is a randomized controlled trial study to measure the effectiveness of a secondary prevention program, called Hastiin Bidziil (Strong Man), aimed at reducing substance use among Native American Indian (AI) men ages 18-26.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as American Indian
* Self-identify as a man
* Age 18-26 years at time of enrollment
* Screen positive for at least moderate risk on any substance, except for tobacco use only
* Reside within ~60 miles of a study community (Fort Defiance, AZ; Chinle, AZ)

Exclusion Criteria:

* Any condition that would affect successful participation (e.g., planned move)
* Profound disability that limits the ability to participate in assessments or interventions
* Participated in the preliminary phase of this study to adapt CETA for this project

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This is a program for people who self-identify as men
Enrollment: 160 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of days of substance sse as assessed by Time Line Follow-back | 6-months post baseline
  Number of days of substance use over the previous month measured at 6-months post baseline using Timeline Follow-Back (TLFB)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Richards, PhD, Principal Investigator — Johns Hopkins University; Jerreed D Ivanich, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Navajo Nation Center for Indigenous Health - Chinle, Chinle, Arizona
  - Navajo Nation Center for Indigenous Health - Fort Defiance, Fort Defiance, Arizona

IPD SHARING:
Plan to Share IPD: No